CLINICAL TRIAL: NCT05795374
Title: Nutritional and Functional Assessment of Patients Undergoing Surgery Due to Gastrointestinal Cancer (NUFAGI): a Prospective Cohort Study.
Brief Title: Nutritional and Functional Assessment of Patients Undergoing Surgery Due to Gastrointestinal Cancer (NUFAGI).
Acronym: NUFAGI
Status: Completed | Type: Observational
Sponsor: Maximos Frountzas (Other)
Responsible Party: Sponsor-Investigator, Maximos Frountzas, Study Coordinator, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Other Study IDs: NUFAGI 2022
Record Dates: First submitted 2023-03-05; First posted 2023-04-03 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Gastrointestinal Cancer
Keywords: nutritional status; functional status; gastrointestinal cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and adipose tissue.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several patients that suffer from gastrointestinal (GI) cancer are characterized by malnutrition and impairment of their functional status. The aim of the present study is to evaluate the nutritional condition of patients undergoing surgery due to GI cancer and compare it with their functional status. All consecutive patients with esophageal, gastric, colorectal, hepatocellular, pancreatic and biliary cancer, that underwent a surgical operation will be included. Demographic characteristics, nutritional assessment and anthropometric measurements of the patients will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a surgical operation due to esophageal, gastric, colorectal, hepatocellular, pancreatic and biliary cancer.

Exclusion Criteria:

* Under 18 years old or above 99 years old.
* Surgery due to benign conditions.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with esophageal, gastric, colorectal, hepatocellular, pancreatic and biliary cancer, that underwent a surgical operation.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity. | 30 days
  Complications after surgery.

SECONDARY OUTCOMES:
Mortality. | 30 days
  Number of deaths.
Disease stage | 1 month
  TNM after histological examination
Recurrence | 1 year
  Disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos G Toutouzas, MD PhD, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Hippocration General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pathirana AK, Lokunarangoda N, Ranathunga I, Santharaj WS, Ekanayake R, Jayawardena R. Prevalence of hospital malnutrition among cardiac patients: results from six nutrition screening tools. Springerplus. 2014 Aug 7;3:412. doi: 10.1186/2193-1801-3-412. eCollection 2014. PMID 25143874
- [Background] Pirlich M, Schutz T, Norman K, Gastell S, Lubke HJ, Bischoff SC, Bolder U, Frieling T, Guldenzoph H, Hahn K, Jauch KW, Schindler K, Stein J, Volkert D, Weimann A, Werner H, Wolf C, Zurcher G, Bauer P, Lochs H. The German hospital malnutrition study. Clin Nutr. 2006 Aug;25(4):563-72. doi: 10.1016/j.clnu.2006.03.005. Epub 2006 May 15. PMID 16698132
- [Background] Huhmann MB, Cunningham RS. Importance of nutritional screening in treatment of cancer-related weight loss. Lancet Oncol. 2005 May;6(5):334-43. doi: 10.1016/S1470-2045(05)70170-4. PMID 15863382
- [Background] Gomes de Lima KV, Maio R. Nutritional status, systemic inflammation and prognosis of patients with gastrointestinal cancer. Nutr Hosp. 2012 May-Jun;27(3):707-14. doi: 10.3305/nh/2012.27.3.5567. PMID 23114934
- [Background] Leandro-Merhi VA, de Aquino JL. Determinants of malnutrition and post-operative complications in hospitalized surgical patients. J Health Popul Nutr. 2014 Sep;32(3):400-10. PMID 25395903